CLINICAL TRIAL: NCT06054100
Title: The Effect of Colchicine on Inflammation in Acute Coronary Syndrome Patients
Brief Title: The Effect of Colchicine on Inflammation in ACS Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanan ahmed, Principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2511
Record Dates: First submitted 2020-02-22; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Acute Coronary Syndrome; STEMI
Keywords: Colchicine; Inflammation; ACS; STEMI; Atherosclerosis
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Inflammation; Atherosclerosis | interventions — Colchicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Electrocardiography parameters assessors and clinical laboratory technicians were masked to the study patient group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine group (Experimental): Colchicine group, Colchicine oral tablets, loading dose 1mg every 12 hrs for 1 day, followed by 0.5 mg BID for 3 months
  Interventions: Drug: Colchicine Tablets
- STEMI standard treatment group (No Intervention): Control group, STEMI standard treatment only

INTERVENTIONS:
Drug: Colchicine Tablets — Colchicine oral tablets loading dose of 1mg every 12 hrs for 1 day, followed by 0.5 mg BID for 3 months
  Other Names: Colchicine
  Arms: Colchicine group

SUMMARY:
This study will evaluate whether the anti-inflammatory effect of colchicine is beneficial in ACS patients

DETAILED DESCRIPTION:
This study will evaluate the effect of colchicine on inflammation, cardiac remodeling, and atherosclerotic risk in STEMI patients through the assessment of the IL-1β, sST2, and lipid profile parameters as well as to examine the drug safety and tolerability in these patients.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* >18 yrs
* STEMI patients who were successfully treated with PCI.

Exclusion Criteria:

* Pregnant or breast-feeding women or women of childbearing potential.
* Active inflammatory, known malignancy, infectious diseases or current treatment with corticosteroids or anti inflammatory agents.
* Known hypersensitivity to colchicine or current chronic treatment with colchicine.
* Severe renal failure (estimated creatinine clearance <30ml/min) or hepatic failure (Child Pugh score B or C )
* Cardiac arrest, ventricular fibrillation, cardiogenic shock or previous myocardial infarction.
* Patients using the following agents: Strong CYP3A4 inhibitors (ritonavir, clarithromycin, ketoconazole, voriconazole, itraconazole), intermediate CYP3A4 inhibitors (aprepitant, diltiazem, erythromycin, fluconazole, verapamil), P-gp inhibitor (amiodarone, clarithromycin, erythromycin, azithromycin, ranolazine, verapamil, ketoconazole, itraconazole) and grape fruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Effect of colchicine therapy on sST2 levels in ACS patients | 3 months
  sST2 level in pg/ml is measured using ELISA method before PCI and after 3 months

SECONDARY OUTCOMES:
Effect of colchicine therapy on occurrence of ischemic events in ACS patients | 3 months
  Effect of colchicine on the occurrence of major adverse cardiovascular events (MACE) during the study period
Change in left ventricular ejection fraction | 3 months
  Effect of colchicine therapy on left ventricular ejection fraction percentage (%)
Change in serum levels of IL-1beta | 3 months
  Effect of colchicine therapy on the change in IL-1beta serum levels in pg/L
Lipid profile parameters and TG/HDL-C ratio | 3 months
  Effect of colchicine therapy on the change in lipid profile parameters and TG/HDL-C ratio

CONTACTS AND LOCATIONS:
Overall Officials: Marwa A Ahmed, Phd, Study Director — Faculty of Pharmacy, Ain Shams University; Lamia El Wakeel, Phd, Study Director — Faculty of Pharmacy, Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassanain HA, El Wakeel LM, Khorshid H, Ahmed MA. Colchicine effect on biomarkers of cardiac remodelling and atherosclerosis in ST-elevation myocardial infarction: A randomized controlled trial. Br J Clin Pharmacol. 2025 Feb;91(2):427-438. doi: 10.1111/bcp.16270. Epub 2024 Oct 2. PMID 39359014